CLINICAL TRIAL: NCT04773808
Title: Implementation of a Comprehensive Multi-level Molecular Strategy for the Identification of Genetic Alterations in Pediatric Solid Tumors Aimed at Achieving a Personalized Approach to the Patient
Brief Title: Molecular Characterization of Genetic Alterations in Pediatric Solid Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Council of Scientific and Technical Research, Argentina (Other Government)
Responsible Party: Principal Investigator, Maria Victoria Preciado, Director of Multidisciplinary Institute for Research of Pediatric Pathologies, National Council of Scientific and Technical Research, Argentina
Other Study IDs: Solid Tumors 2020
Record Dates: First submitted 2021-02-19; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Pediatric Solid Tumors
Keywords: pediatric solid tumor; molecular marker; molecular tumor profile; tailored therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: In Argentina, central nervous system (CNS) solid tumors (19%) and non-CNS solid tumors (25%) account for 44% of pediatric tumors. The new World Health organization (WHO) 2016 classification, which includes genomic characterization, comprises more than 100 CNS tumor entities and subclasses. In children, glial lineage tumors (gliomas) are the most frequent and comprise astrocytomas, ependymomas and oligodendroglioma, while embryonal CNS tumors are a heterogeneous group of WHO grade IV tumors. Pediatric soft tissue tumors (STT) present difficulties for accurate diagnosis since their morphological and immunophenotypic features overlap among the different histological patterns.

The emergence of new molecular techniques has generated a great advance in the field of solid tumors, particularly in the molecular definition of groups of patients. This fact makes tailor-made treatment feasible, according to the biology of the tumor.

In particular, in children, the identification of treatment targets is especially important since it may avoid unnecessary sequel in a growing child. This project allows the articulation between basic and clinical research groups, thus consolidating the objective of basic translational research and generating both clinical and basic knowledge about the pathogenesis of pediatric solid tumors in our country.

Aim: To standardize and implement a comprehensive multi-level molecular strategy, using medium and high complexity techniques, for the detection of molecular alterations in primary pediatric solid tumors (neuroblastoma, rhabdomyosarcoma, Ewing sarcoma family tumors, soft tissue sarcomas and CNS tumors (gliomas and embryonal)), that can be applied to the diagnosis, prognosis and/or use of targeted therapies against molecular targets in order to provide a tailored therapeutic opportunity.

Material and methods: Pediatric cases of solid tumors will be enrolled prospectively. Based on the statistics of the participating centers, 100 samples will be included. From each case, a formalin fixed biopsy will be available and when possible, a fragment will also be preserved at -70ºC. Clinical and follow-up data will be obtained from the clinical records.

The methodological approaches include: 1) Immunohistochemical detection of tumor lineage determinant markers, some of them with predictive value. 2) FISH (fluorescence in situ hybridization) with break-apart strategy for genes involved in recurrent chromosomal translocations and locus-specific design probes for other unbalanced structural chromosomal structural alterations (amplifications and deletions of genes or chromosomal segments). 3) Real time (RT)-polymerase chain reaction (PCR) detection of fusion transcripts resulting from chromosomal translocations. 4) Quantitative polymerase chain reaction (qPCR) and Sanger sequencing analysis of single nucleotide polymorphisms (SNPs) as targets for therapy. 5) Sanger sequencing analysis of fusions, ins/del as a complement to RT-PCR or FISH (fluorescence in situ hybridization), 6) Next Generation Sequencing (NGS) with a specific and customized panel containing all necessary genes to define a tumor´s genomic mutation profile for diagnosis, risk stratification and prognosis of pediatric tumors. However, NGS sequencing will only be applied in those cases which could not be resolved with the previous strategies or cases with poor evolution

Based on the above analyses, an integrated analysis algorithm will be developed according to WHO recommendations, but adapted to the facilities of the institution. Molecular findings will be correlated with clinical and histological data

ELIGIBILITY:
Inclusion Criteria:

1. Must have a suspected or known diagnosis of neuroblastoma, rhabdomyosarcoma, Ewing sarcoma family tumors, soft tissue sarcomas and CNS tumors (gliomas and embryonal) based on the initial diagnostic workup and evidence of gross disease amenable to excision. Specimens may be collected at some or all of the following time points: initial biopsy, tumor resection and at time of possible relapse.
2. The patient or his/her legal guardian, as appropriate, must provide written informed consent within 30 days of the removal of the first collection of tissue sample for this protocol.
3. The patient is being seen at Hospital de Niños R Gutierrez or at a collaborating institution.
4. Patients must be less than or equal to 18 years old at the time of enrollment.

Exclusion Criteria:

1. No access to the tumor tissue sample.
2. written informed consent is not obtained.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients identified at Hospital de Niños R Gutierrez and collaborating institutions with a suspected or known diagnosis of neuroblastoma, rhabdomyosarcoma, Ewing sarcoma family tumors, soft tissue sarcomas and CNS tumors (gliomas and embryonal), based on initial diagnosis through clinical examination, laboratory testing and images of a mass ameneable to excision
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
molecular profiling of solid tumors | 5 years
  Perform molecular identification of genetic alterations in neuroblastoma, rhabdomyosarcoma, Ewing sarcoma family tumors, soft tissue sarcomas and CNS tumors (gliomas and embryonal)

SECONDARY OUTCOMES:
molecular markers analysis vby immunohistochemistry | 5 years
  1) Perform immunohistochemical analysis of tumor lineage determinant markers some of them with predictive value
molecular markers analysis by fluorescence in situ hybridization | 5 years
  2) Perform FISH (fluorescence in situ hybridization) analysis of recurrent chromosomal translocations and structural chromosomal alterations
molecular markers analysis by gene amplification | 5 years
  3) Perform RT-qPCR analysis for gene translocations and qPCR analysis for reported SNPs
molecular markers analysis by sequencing | 5 years
  4) Perform complementary Sanger sequencing analysis for SNPs and translocations of unresolved cases
molecular markers analysis by Next Generation Sequencing | 5 years
  5) Perform Next Generation Sequencing (NGS) with a specific and customized panel to define a tumor genomic mutation profile important in the diagnosis, risk stratification and prognosis

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Victoria Preciado, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided